CLINICAL TRIAL: NCT00439816
Title: Veteran Preference For Group Visits and Its Effect on Hypertension Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LIP 82-003; HR 11260
Record Dates: First submitted 2007-02-22; First posted 2007-02-26 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-11

CONDITIONS: Hypertension; Blood Pressure
Keywords: Hypertension Outcomes; Health Outcomes; Outpatient; Racial Preference; Blood Pressure Control; Clinical Trial; Intervention; Lifestyle modifications; Ethnic Differences; Randomized
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Behavioral: Group Visits

INTERVENTIONS:
Behavioral: Group Visits

SUMMARY:
To determine racial/ethnic differences in preference for group visits in veterans with poorly controlled hypertension (State 2 hypertension) and determine the effect of group visits on health outcomes among veterans with poorly controlled hypertension.

DETAILED DESCRIPTION:
Research Design: Randomized clinical trial to assess veterans� preference for group visits and the effect of group visits on hypertension outcomes. Hypertension affects close to 50 million persons in the U.S., with prevalence, severity, and impact being increased in non-white Americans 1.Despite recent clinical trials associating successful antihypertensive therapy with reductions in stroke incidence, myocardial infarction, and heart failure, control rates remain below the Healthy People 2010 goal of 50%. The importance of blood pressure control is recognized within the VA as two of the conditions selected for QUERI include ischemic heart disease and congestive heart disease, and blood pressure control is a performance measure for every VAMC 2. Clinical trials have shown that blood pressure control can be achieved in most patients with hypertension 3. When physicians fail to prescribe lifestyle modification, adequate doses of antihypertensive medications, or appropriate drugs, blood pressure control may not be achieved.1 In the course of a 15-30 minute visit with a primary care physician, lifestyle modifications may not be addressed and inertia may prevent rapid adjustments in medication dosages or changes in drug combinations. 4. The outpatient group visit model is an intervention developed by managed care organizations to capitalize on economy of scale. It has significant points of departure from the existing health care delivery system design, which focuses on acute care. The outpatient group visit model also fosters a more collaborative effort between the physician and patient, introduces nurses as knowledgeable team members who can be trusted to communicate important information to patients and between patients and physicians, and promotes peer support among the participating patients. Group visits have proven successful in high health services utilizing elderly patients with one or more chronic illnesses. A one-year study of monthly 2-hour group visits led by a physician and nurse showed significant improvements in care delivery as measured by decreases in emergency room visits, specialty care visits, and hospital readmissions though no change in self-reported health and functional status were realized. 5. Also, patients with type 2 diabetes attending group visits were shown to have increases in quality of life measures, knowledge of type 2 diabetes, and improved metabolic control as compared to patients in usual care. 6. Group visits offer providers more time per visit to address process-of-care indicators and provide patients more time per visit with their primary care physician. The monthly schedule allows for more frequent contacts between the patients and physicians. Providers caring for patients in groups can deliver consistent messages to multiple patients at once. Though monthly primary care visits (in groups) would be an increase from the 4 primary care visits per year presently realized by veterans with hypertension at the Ralph H. Johnson VAMC, the frequency is more consistent with JNC 7 guidelines for monthly visits for follow-up and monitoring after the initiation of antihypertensive therapy. Presently, the average primary care physician at the Charleston VA is scheduled to see 2 patients per hour. Group visits would allow the physician to see 20 patients over 2 hours. While demonstrated feasible and acceptable to elderly, chronically ill managed care populations, and uninsured and underinsured patients with type 2 diabetes, group visits have not been systematically tested in the Veteran�s Health Administration system. Additionally, previous studies have not evaluated patients� acceptance of group visits or their responses to groups according to race/ethnicity. This study seeks to inform whether group visits are acceptable to veterans as a method of health care delivery, regardless of race/ethnicity.

Methods: The study will assess the effect of group visits on hypertension outcomes. Veterans with stage 2 hypertension (systolic blood pressure =160 mmHg or diastolic blood pressure =100 mmHg) will be identified during routine office visits. The primary care physician will explain what group visits are using a standard script then patients will be asked if they are willing to be seen in a group setting. Patients who indicate a willingness to receive care in a group setting will be randomly assigned to either group visits or usual care. Randomization will occur in blocks to insure equal number of subjects by race/ethnicity in each of the two groups (group setting vs. usual care). We will recruit up to 8 VA primary care physicians to participate in this study. Several have already indicated an interest in conducting group visits.

Patient Visit Protocol: Group visits will be co-led by the patients� primary care internal medicine physician and a clinic nurse. Each group visit session will be scheduled for two hours consisting of: 15 minutes for "warm-up" and socialization, 30 minutes for presentation of a health- related topic (facilitated by the physician or another team member with special expertise), 15 minutes for break, during which time the nurse and physician will circulate, attending to individual needs, immunizations, appointment scheduling, and other issues, 15 minutes for questions and answers, 15 minutes for planning the next session, and 30 minutes for one-on-one consultations with the physician. Upon conclusion of the group portion of the visit, patients will have the opportunity to see the physician individually if required. While the group visits are intended to be the main source of medical care, patients who need care in between scheduled group visits, or who have specific medical needs that cannot be accommodated in the group visit (i.e. PAP smears, DRE), will be able to schedule a one-on-one visit with their primary care provider.

ELIGIBILITY:
Inclusion Criteria:

Caucasian and African American men and women, age 21 and older with stage 2 hypertension presently seen in the RHJ VAMC Primary Care.

Exclusion Criteria:

Primary diagnosis of substance abuse or dependence, current pregnancy, dementia, inability to speak English, or controlled psychiatric diagnoses.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2005-02; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Blood pressure control. Medication compliance (as measured by refill histories). Health services utilization patterns (as defined by days in hospital, outpatient visits and urgent care visits).

SECONDARY OUTCOMES:
Acceptability of group visits to White and African American veterans, measured by comparing proportion of those who agreed to participate in groups to those who didn't. The attendance rates by patient race/ethnicity among those assigned to group visits.

CONTACTS AND LOCATIONS:
Overall Officials: Dawn E Clancy, MD, Principal Investigator — Ralph H. Johnson VA Medical Center, Charleston, SC
Locations (1):
- Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina, United States

REFERENCES:
- [Result] Wager KA, Ward DM, Lee FW, White AW, Davis KS, Clancy DE. Physicians, Patients, and EHRs. When it comes to a consultation, is three a crowd? J AHIMA. 2005 Apr;76(4):38-41. No abstract available. PMID 15871467
- [Result] Davis KS, Magruder KM, Lin Y, Powell CK, Clancy DE. Brief report: Trainee provider perceptions of group visits. J Gen Intern Med. 2006 Apr;21(4):357-9. doi: 10.1111/j.1525-1497.2006.00350.x. PMID 16686812